CLINICAL TRIAL: NCT01451671
Title: Prenatal Test for Fetal Aneuploidy Detection
Brief Title: Development of a Prenatal Test for Fetal Aneuploidy Detection
Status: Completed | Type: Observational
Sponsor: Cindy Cisneros (Industry)
Responsible Party: Sponsor-Investigator, Cindy Cisneros, CRA, Roche Sequencing Solutions
Organization: Roche Sequencing Solutions (Industry)
Other Study IDs: TD002
Record Dates: First submitted 2011-10-10; First posted 2011-10-14 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Fetal Complications
Keywords: fetal; aneuploidy; non-invasive; prenatal; cell free DNA
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study to develop and evaluate a blood based prenatal blood test. Pregnant women confirmed to be carrying a fetus with a chromosomal abnormality will be eligible. Subjects will be asked to provide a blood sample and a limited amount of clinical data that will be recorded on a case report form. All samples and clinical data will be stripped of subject identifiers prior to submission to Ariosa.

ELIGIBILITY:
Inclusion Criteria:

* Subject has singleton pregnancy
* Subject is confirmed via invasive testing to be carrying a fetus with a chromosomal abnormality
* Subject is able to provide informed consent
* Subject is ≥ 18 years of age

Exclusion Criteria:

* Subject is pregnant with more than one fetus
* Subject (mother) has a known aneuploidy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women carrying a fetus with an abnormal chromosomal condition that has been confirmed by invasive testing.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2010-11; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Identification of aneuploidy | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Roberts, Study Director — Ariosa Diagnostics
Locations (3):
- United States (3):
  - University of California San Diego, San Diego, California
  - Norton Healthcare, Louisville, Kentucky
  - Medical College of Wisconsin, Milwaukee, Wisconsin